CLINICAL TRIAL: NCT06433258
Title: Implementation and Evaluation of an Evidence-Based, Multilevel Lifestyle Intervention for Underserved and Rural Populations in South Texas: Tu Salud ¡Si Cuenta (TSSC)!
Brief Title: Implementation and Evaluation of an Evidence-Based, Multilevel Lifestyle Intervention for Underserved and Rural Populations in South Texas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Belinda Reininger, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-1025
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cancer Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced TSSC curriculum (Experimental)
  Interventions: Behavioral: Enhanced TSSC curriculum
- Original TSSC curriculum (Active Comparator)
  Interventions: Behavioral: Original TSSC curriculum

INTERVENTIONS:
Behavioral: Enhanced TSSC curriculum — In addition to the original TSSC curriculum participants will also be educated with the enhanced curriculum which includes components related to alcohol and social determinants of health needs) to promote cancer prevention through healthy lifestyles.
  Arms: Enhanced TSSC curriculum
Behavioral: Original TSSC curriculum — Participants will be educated with evidence-based modules focused on topics such as introduction to TSSC, physical activity, fruit and vegetable consumption, reduce sugar intake, diabetes, portion control, cancer, and high blood pressure.These modules are provided by community health workers who have been trained in the contents of the modules, as well as motivational interviewing techniques for delivering the modules.
  Arms: Original TSSC curriculum

SUMMARY:
The purpose of this study is to enhance the current TSSC multilevel intervention delivered in Cameron and Hidalgo counties by adding additional components including an educational module on the risks of alcohol intake and its connection to cancer, as well as developing training and referral systems to address social determinants of health (SDOH) that negatively impact uptake of cancer prevention behaviors.

ELIGIBILITY:
Inclusion Criteria:

* residents of partnering municipalities throughout Cameron and Hidalgo

Exclusion Criteria:

* participated in TSSC before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of participants that show an increase in moderate and vigorous physical activity minutes as assessed by the Physical Activity Questionnaire | Baseline , 6 month follow up , 9 month month follow up
Change in percentage of participants that report increase in fruit and vegetable intake as assessed by the Nutritious Eating Questionnaire | Baseline , 6 month follow up , 9 month month follow up
Change in percentage of participants that report a reduced quantity of alcohol intake as assessed by a questionnaire | Baseline , 6 month follow up , 9 month month follow up
Change in percentage of participants that report a reduced frequency of alcohol intake as assessed by a questionnaire | Baseline , 6 month follow up , 9 month month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Reininger, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No